CLINICAL TRIAL: NCT03327168
Title: Adenosine and A2a Receptors in Human Brown Adipose Tissue (AdenoBAT)
Brief Title: Adenosine and A2A Receptors in Human Brown Adipose Tissue
Acronym: AdenoBAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Bonn (Other)
Responsible Party: Principal Investigator, Kirsi Virtanen, Adjunct Professor, Turku University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: T201/2015
Record Dates: First submitted 2017-09-28; First posted 2017-10-31 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Obesity
Keywords: Adipose Tissue, Brown
MeSH Terms: conditions — Obesity | interventions — Adenosine

STUDY DESIGN:
Intervention Model Description: Each subject participates in PET/CT scans in room temperature conditions, during cold exposure and during i.v. infusion of adenosine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adenosine (Active Comparator): Perfusion is measured using PET/CT during intravenous infusion (0.14 mg/kg/min) of adenosine.
  Interventions: Drug: Adenosine
- Room temperature (No Intervention): Perfusion and A2A receptor density is measured using PET/CT in resting room temperature conditions.
- Cold exposure (Experimental): Perfusion and A2A receptor density is measured using PET/CT during controlled cold exposure.
  Interventions: Other: Cold exposure

INTERVENTIONS:
Drug: Adenosine — Intravenous infusion of adenosine (0.14 mg/kg) is administered for 5 minutes during PET/CT scan.
  Other Names: Adenocor
  Arms: Adenosine
Other: Cold exposure — Controlled cold exposure is performed before and during PET/CT scan.
  Arms: Cold exposure

SUMMARY:
This study investigates the significance of adenosine and A2A receptors in human brown adipose tissue (BAT) in vivo. Using positron emission tomography (PET), perfusion and the density of A2A receptors will be measured in supraclavicular BAT and other tissues in healthy men. The investigators hypothesize, that adenosine can activate BAT, and that adenosine A2A receptor density changes when BAT is activated by cold exposure.

Understanding the mechanisms of BAT activation and the role of endocannabinoids in humans is important and beneficial in fighting against the epidemic of obesity and diabetes.

DETAILED DESCRIPTION:
Adenosine is a purine nucleoside released locally in BAT when noradrenaline and ATP are released from sympathetic nerves. Recently it was found that adenosine activates murine and human brown adipocytes, and recruits beiging of white fat via adenosine A2A receptors (A2AR). Furthermore, studies with mice have shown improvements in glucose homeostasis after administration of A2AR agonists.

In this study the investigators use the PET radiotracer [15O]-H2O to quantify perfusion of BAT, white adipose tissue (WAT) and muscle in three conditions: room temperature, cold exposure and intravenous infusion of adenosine. Another PET radiotracer [11C]TMSX is used to quantify adenosine A2A receptor density of BAT, WAT and muscle in room temperature and during cold exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Male sex
2. BMI 20 - 28 kg/m2
3. Age: 18- 40 years
4. Normal OGTT
5. Healthy, no regular medication

Exclusion Criteria:

1. BMI < 20 kg/m2 or BMI > 28 kg/m2
2. Low or high blood pressure
3. Asthma or other obstructive lung disease
4. Sick sinus syndrome, prolonged QT-interval, or any heart disease
5. Any chronic disease that could affect the study outcome, including diabetes
6. Mental disorder or poor compliance
7. Eating disorder or excessive use of alcohol, tobacco smoking or drug use
8. Past dose of radiation
9. Any other condition that in the opinion of the investigator could create a hazard to the subject safety, endanger the study procedures or interfere with the interpretation of study results

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
BAT perfusion | Effect within 10 minutes
  Perfusion of BAT with [15O]-H2O PET-CT
A2A receptor density in BAT | Effect within 3 hours
  Density of A2A receptors in BAT measured with [11C]-TMSX PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Kirsi A Virtanen, MD, PhD, Principal Investigator — Turku University Hospital

IPD SHARING:
Plan to Share IPD: No